CLINICAL TRIAL: NCT07151833
Title: Efficacy of GlucoBites Functional Cookies Containing Gynura Procumbens on Glycemic Control, Insulin Resistance, and Prevention of Diabetic Foot Ulcer Risk in Patients With Type 2 Diabetes Mellitus: A Randomized Controlled Trial
Brief Title: GlucoBites Cookies (Gynura Procumbens) for Glycemic Control and Prevention of Diabetic Foot Ulcer Risk in Type 2 Diabetes
Acronym: GlucoBites
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Andina Setyawati (Other)
Responsible Party: Sponsor-Investigator, Andina Setyawati, Principal Investigator, Hasanuddin University
Organization: Hasanuddin University (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: GlucoBites-DM2-2025; 02209/UN4.22/PT.01.03/2025 (Other Grant/Funding Number: BIMA Research Grant 2025)
Record Dates: First submitted 2025-08-22; First posted 2025-09-03 (Actual); Last update posted 2025-09-03 (Actual); Status verified 2025-09

CONDITIONS: Type 2 Diabetes Mellitus; Diabetic Neuropathy
Keywords: Diabetes Mellitus Type 2; Functional Food; Gynura procumbens; Glycemic Control; Insulin Resistance; Diabetic Foot Ulcer Prevention
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Diabetic Neuropathies; Insulin Resistance

STUDY DESIGN:
Intervention Model Description: This randomized controlled trial uses a parallel assignment model with two study arms. Participants will be randomly allocated to either the intervention group receiving GlucoBites functional cookies containing Gynura procumbens or the control group receiving standard diabetes care. Both groups will be followed simultaneously for 12 weeks.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Participants in both arms receive visually identical cookies. The experimental cookies contain Gynura procumbens extract, while the control cookies do not. Packaging, appearance, weight, and flavor are matched. Randomization codes are held by an independent pharmacist/allocator; care providers and outcomes assessors are blinded to group assignment. Unblinding will occur only after database lock or for safety reasons.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Cookies (without Gynura procumbens) (Placebo Comparator): Participants receive 4 cookies per day for 12 weeks. The cookies are identical in packaging, size, weight, and flavor but do not contain Gynura procumbens.
  Interventions: Dietary Supplement: Control Cookies (without Gynura procumbens)
- GlucoBites (with Gynura procumbens) (Experimental): Participants receive 4 cookies per day for 12 weeks. The cookies contain standardized Gynura procumbens extract.
  Interventions: Dietary Supplement: GlucoBites (with Gynura procumbens)

INTERVENTIONS:
Dietary Supplement: GlucoBites (with Gynura procumbens) — Participants receive 4 cookies per day for 12 weeks. The cookies contain standardized Gynura procumbens extract.
  Other Names: Functional Cookies with Gynura procumbens
  Arms: GlucoBites (with Gynura procumbens)
Dietary Supplement: Control Cookies (without Gynura procumbens) — Participants consume 4 cookies per day for 12 weeks. The cookies are identical in packaging, size, weight, and flavor to the GlucoBites cookies but do not contain Gynura procumbens.
  Other Names: Placebo cookies
  Arms: Control Cookies (without Gynura procumbens)

SUMMARY:
The goal of this randomized controlled trial is to learn if GlucoBites functional cookies containing Gynura procumbens can help improve blood sugar control and lower the risk of diabetic foot ulcers in adults with type 2 diabetes.

The main questions are:

* Do GlucoBites cookies lower fasting blood glucose and HbA1c?
* Do GlucoBites cookies improve insulin resistance and vascular health?
* Can GlucoBites reduce early signs that may lead to diabetic foot ulcers?

Researchers will compare:

* Intervention group: participants will eat 4 GlucoBites cookies every day for 12 weeks.
* Control group: participants will continue standard diabetes care without GlucoBites.

Participants will:

* Visit the community health center for blood tests and foot health checks.
* Be monitored for blood sugar, insulin resistance, lipid profile, and vascular function.
* Be assessed for early risk of diabetic foot ulcer development.

This study will help determine if a functional food innovation can support diabetes care and prevent complications.

DETAILED DESCRIPTION:
Type 2 diabetes mellitus is a chronic condition associated with serious complications, including neuropathy and diabetic foot ulcers. Many people in Indonesia still struggle with poor blood sugar control despite standard treatments. This highlights the need for safe, affordable, and culturally acceptable nutritional strategies.

This study is testing GlucoBites, a functional cookie made with Gynura procumbens, a traditional medicinal plant with potential glucose-lowering and vascular protective properties. Researchers want to see if adding GlucoBites to daily care can improve blood sugar control and reduce early risk factors linked to diabetic foot ulcer development.

The study will help determine whether functional food innovation can be integrated into community-based diabetes management and offer a preventive approach to reduce long-term complications.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 20-70 years.
* Diagnosed with type 2 diabetes mellitus (T2DM) based on ADA criteria.
* HbA1c ≥ 7%.
* At risk of diabetic foot ulcer (ABI < 0.9 or early neuropathy signs).
* Willing to consume study cookies and comply with study protocol.
* Provided written informed consent.

Exclusion Criteria:

* Current use of herbal supplements or functional foods containing Gynura procumbens.
* Presence of active diabetic foot ulcer or severe infection.
* Severe cardiovascular, renal (eGFR < 30 mL/min/1.73 m²), or hepatic impairment.
* Pregnancy or breastfeeding.
* Known allergy to ingredients in study cookies.
* Participation in another clinical trial within the last 3 months.

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 126 (Estimated)
Dates: Start 2025-09-20 (Estimated); Primary Completion 2025-12-20 (Estimated); Study Completion 2026-01-20 (Estimated)

PRIMARY OUTCOMES:
Fasting Blood Glucose (FBG) | Baseline and 12 weeks after intervention
  Fasting blood glucose (FBG, mg/dL) measured from venous blood after 8-10 hours of fasting using standardized laboratory methods. The primary endpoint is the change from baseline to Week 12, comparing the GlucoBites group (with Gynura procumbens) and the control group (without Gynura procumbens).
Change in HOMA-IR | Baseline and 12 weeks after intervention
  Homeostatic Model Assessment of Insulin Resistance (HOMA-IR) calculated from fasting glucose (mg/dL) and fasting insulin (µIU/mL) using the formula: [fasting insulin × fasting glucose / 405]. The endpoint is the change in HOMA-IR from baseline to Week 12, comparing the GlucoBites group (with Gynura procumbens) and the control group (without Gynura procumbens).
MMP-9/TIMP-1 Ratio | Baseline and 12 weeks after intervention
  The ratio of matrix metalloproteinase-9 (MMP-9) to tissue inhibitor of metalloproteinase-1 (TIMP-1) in serum, quantified using ELISA. The ratio is calculated by dividing MMP-9 (ng/mL) by TIMP-1 (ng/mL). The endpoint is the change in MMP-9/TIMP-1 ratio from baseline to Week 12, comparing the GlucoBites group (with Gynura procumbens) and the control group (without Gynura procumbens).
Ankle-Brachial Index (ABI) | Baseline and 12 weeks after intervention
  The ankle-brachial index (ABI) is calculated as the ratio of systolic blood pressure measured at the ankle to systolic blood pressure measured at the brachial artery. Measurements are obtained using a handheld Doppler device. ABI will be used as an indicator of peripheral vascular function and early risk of diabetic foot ulcer. The endpoint is the change in ABI from baseline to Week 12, comparing the GlucoBites group (with Gynura procumbens) and the control group (without Gynura procumbens).

CONTACTS AND LOCATIONS:
Locations (1):
- Public Health Centre of Campagaloe, Bantaeng, South Sulawesi, Indonesia

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data (IPD) underlying the published results will be made available in anonymized form. The data will be accessible upon reasonable request to the corresponding investigator after publication, in accordance with ethical approval and institutional policies
Supporting Information: Study Protocol, SAP, ICF
Time Frame: IPD and supporting documents (study protocol, statistical analysis plan, and informed consent form) will be available within 6 months after publication of the main results and will remain available for 5 years
Access Criteria: De-identified individual participant data (IPD) and supporting documents will be available to qualified researchers for academic and scientific purposes. Access will be granted upon reasonable request to the sponsor or principal investigator, subject to approval of a data use agreement

REFERENCES:
- See also: Original research article reporting the antidiabetic effects of Gynura procumbens on pancreatic histopathology via caspase family expression in diabetic rat models, published in the Journal of Pharmacy & Pharmacognosy Research (2025). — https://jppres.com/jppres/pdf/vol13/jppres24.2112_13.3.836.pdf